CLINICAL TRIAL: NCT03632785
Title: Laboratory Implications of Non Obstructive Atherosclerotic Plaques Identified by Multiple Detector Coronary Angiotomography
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Jose Carlos Nicolau, Professor, PhD., University of Sao Paulo
Other Study IDs: FAPESP 2014/01021-4 - Subp. 1
Record Dates: First submitted 2018-08-05; First posted 2018-08-15 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Discrete Coronary Artery Stenosis; Coronary Angiography of Multiple Detectors; Platelet Aggregation, Spontaneous; Cardiovascular Risk Factor
Keywords: Platelet; Coronary stenosis; Coronary angiography
MeSH Terms: conditions — Platelet Aggregation, Spontaneous; Coronary Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Approximately 50% of coronary events occur in previously asymptomatic patients. Thus, the early detection of the individuals at higher risk became an important research target within the current cardiology. The various clinical scores used present a predictive accuracy for ischemic events, evaluated by the ROC curve, which ranges from 0.73 to 0, 79. Therefore, the introduction of new non-invasive techniques for the detection of atherosclerosis aims to allow a more adequate classification of risk. The development of radiological techniques, fundamentally coronary angiotomography of multiple detectors (CAMD) and electron beam computed tomography-EBCT‖, demonstrated that the degree of coronary calcification correlates with endothelial lesion and individual prognosis in the long term. Notably, the calcium score has a weak correlation with the severity of coronary stenosis per se, possibly due to variations in arterial remodeling due to coronary calcification. On the other hand, the CAMD allows the detection of a small magnitude atheromatous disease, not diagnosed clinically, nor by tests provoking ischemia, or even by coronary catheterization.

The clinical relevance of the small magnitude atheromatous disease diagnosed by the ACMD and its correlation with plaque vulnerability markers, mainly platelet aggregation, vascular reactivity, and inflammation are still not well determined.

This is a case and control study and we will enrolled 90 patients with low and medium risk of cardiovascular event whose cases should present discrete plaques in the CAMD e controls should present none plaque in coronary stenosis

DETAILED DESCRIPTION:
Coronary atherosclerotic disease often begins in the transition from childhood to adolescence, progressing slowly and quietly. Its clinical manifestation occurs in the majority of cases from the 4th decade of life. However, it is important to remember that necropsy studies conducted in the 1970s identified the presence of non-obstructive atherosclerotic plaques in the aorta of individuals from the second decade of life.

From its first description to the present day, the subject has been deeply studied, providing reliable information on several mechanisms involved in atherogenesis, disease progression and plaque unstabilization, which may occur in a silent manner or lead to a clinical picture of unstable myocardial ischemic syndrome (UMIS). In this period, classic risk factors for coronary artery disease (age, sex, diabetes mellitus, systemic arterial hypertension, hypercholesterolemia and smoking, among others) were described, and risk scores were developed that aid in the individual prediction of the probability of disease manifestation coronary artery disease (CAD).

The most widespread of these scores is that developed from the population of Framingham, which was started in the United States of the same name after 1948. Subjects with no evidence of cardiovascular disease were followed prospectively with biannual evaluations. The data obtained allowed the elaboration of an algorithm of prediction of individual risk that is included in the most recent recommendations of evaluation of cardiovascular risk.

However, these traditional clinical assessment scores tend to underestimate cardiovascular risk in some populations, especially in women and young individuals. In the global population, the various clinical scores used have a predictive accuracy for ischemic events, as assessed by the ROC (Receiver Operating Characteristic) curve, ranging from 0.73 to 0.79.

In this way, the concept of "detection interval" is proposed. Defined by the difference between cases of coronary disease or cardiovascular events detected and the actual total prevalence of atherosclerotic disease in the population, such detection interval opens a new field for the introduction of new non-invasive atherosclerosis investigation techniques.

Taking into account that approximately 50% of coronary events occur in previously asymptomatic patients, the early detection of these individuals at greater risk has become an important research target within the current cardiology.

More recently, the development of radiologic techniques, fundamentally coronary angiography of multiple detectors (CAMD) and electron beam computed tomography (EBCT), have demonstrated that the degree of coronary calcification correlates with endothelial lesion and individual prognosis in the long term, allowing to refine the clinical classification of a patient's risk for a greater or lesser chance of fatal and non-fatal events. Notably, the calcium score has a weak correlation with the severity of coronary stenosis per se, possibly due to variations in the arterial remodeling due to coronary calcification.

On the other hand, calcification of the coronary arteries is known to be associated with lower myocardial blood flow even in the absence of significant stenosis. This means that calcification is not merely a marker of obstructive coronary disease and may predispose patients to myocardial ischemia by mechanisms other than those traditionally known and may therefore be a marker of endothelial dysfunction.

On the other hand, the application of CAMD allowed the detection of a small magnitude atheromatosis , not diagnosed clinically by the tests provoking ischemia or even by contrast-enhanced coronary angiography. The clinical relevance of these alterations, evaluated by their correlation with the presence of plaque vulnerability markers, mainly platelet aggregation, vascular reactivity, and inflammation, is still very little studied, being the main objective of this study.

ELIGIBILITY:
Inclusion Criteria:

* Low or Medium Risk of cardiovascular disease assessed by the Framingham criteria;
* That agrees to sign the Consent Form;
* Absence of known atherosclerotic disease;
* Patients in the case group should additionally present discrete plaques (s) evaluated by coronary angiotomography of multiple detectors (CAMD). Patients in the control group should be absent from any coronary atherosclerotic process to CAMD.

Exclusion Criteria:

* Known atherosclerotic disease manifest;
* Previous acute coronary syndrome (ACS);
* Use of antiplatelet agents and / or anticoagulants;
* Use of NSAIDs and/or corticosteroids
* Known platelet dysfunction or platelets <100,000 / μL or> 450,000 / μL
* Hematocrit <33% and > 52%
* Hematological diseases;
* Liver disease;
* Known malignant neoplasm;
* Refusal to sign free and informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years, male and female with low and medium risk of cardiovascular disease without atherosclerotic disease manifest.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation by VerifyNow System - P2Y12® | 1 day
  Comparing platelet aggregation by VerifyNow System - P2Y12® (An equipment from Accriva Diagnostics that evaluates platelet aggregation) in case and control groups.

SECONDARY OUTCOMES:
Platelet aggregation by Multiplate-ADP®, Multiplate-ASPI® | 1day
  Comparing platelet aggregation by Adenosine Diphosphate pathway (ADP test) and by Arachidonic Acid pathway (ASPI test). Theses methods will be analyzed in case and control groups.
Endothelial function | 1 day
  Comparing endothelial function by ENDOPAT 2000 method (is the leading medical device for noninvasive endothelial function assessment. It was developed and is distributed by Itamar Medical, Caesarea, Israel) in case and control groups
Platelet-reticulated | 1day
  comparing platelet-reticulated analysis in the case and control groups;
Inflammatory activity | 1day
  Comparing the inflammatory activity by Interleukin 6 (IL-6) and by Ultra-Sensitive C-Reactive Protein (us-CRP) in the case and control groups

OTHER OUTCOMES:
Genetic polymorphisms | 1day
  Comparing the presence of genetic polymorphisms in the case and control groups;
Transport of lipids to HDL | 1 day
  Comparing Transport of lipids to HDL in the case and control group
Correlate results | through study completion, an average of 1 year
  Correlate platelet aggregability with inflammatory markers and presence of polymorphisms; and. Comparing platelet aggregation among patients with or without calcium (in the ACMD) of the case group
Comparing platelet aggregation in subgroups | through study completion, an average of 1 year
  Comparing platelet aggregation in the case and control groups in the following subgroups:
  * Diabetics and non-diabetics;
  * Elderly (≥65 years) and not elderly;
  * Feminine and masculine genres;
  * With renal dysfunction (Clearance Creatinine <60) and without renal dysfunction;
  * With statin and without statin.
  * Obese (IMC≥30) and non-obese
  * Smoking / non-smoking
Global Risk Score | through study completion, an average of 1 year
  Comparing Global Risk Score (global risk of coronary heart disease - is a calculation of the absolute risk of having a coronary heart disease event in 10 years. Some variables are analyzed: Age (40-79 years), Gender (male or female), Total cholesterol (130-320mg/dL), HDL cholesterol(20-100mg/dL), Systolic blood pressure (90-200mmHg), Diastolic blood pressure (30-140mmHg), Treated for high blood pressure (Yes ou Not), Diabetes (Yes or Not) and Smoker (Yes or Not). After calculation we have a final number and its respective risk (%) of developing cardiovascular disease. With this, we classify the patient in Low risk(< 5% to have coronary disease in 10 years), Moderate Risk ( Men ≥ 5% e ≤ 20% and Woman ≥ 5% e ≤ 10%) and High risk ( Men >20% and Woman > 10%). We will compare this Global Risk Score in case and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- José Carlos Nicolau, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavi S, Bae JH, Rihal CS, Prasad A, Barsness GW, Lennon RJ, Holmes DR Jr, Lerman A. Segmental coronary endothelial dysfunction in patients with minimal atherosclerosis is associated with necrotic core plaques. Heart. 2009 Sep;95(18):1525-30. doi: 10.1136/hrt.2009.166017. Epub 2009 Jun 3. PMID 19497916
- [Result] Deanfield JE, Halcox JP, Rabelink TJ. Endothelial function and dysfunction: testing and clinical relevance. Circulation. 2007 Mar 13;115(10):1285-95. doi: 10.1161/CIRCULATIONAHA.106.652859. No abstract available. PMID 17353456
- [Result] Ross R, Harker L. Hyperlipidemia and atherosclerosis. Science. 1976 Sep 17;193(4258):1094-100. doi: 10.1126/science.822515.
- [Result] Wilson PW, D'Agostino RB, Levy D, Belanger AM, Silbershatz H, Kannel WB. Prediction of coronary heart disease using risk factor categories. Circulation. 1998 May 12;97(18):1837-47. doi: 10.1161/01.cir.97.18.1837. PMID 9603539
- [Result] Greenland P, Alpert JS, Beller GA, Benjamin EJ, Budoff MJ, Fayad ZA, Foster E, Hlatky MA, Hodgson JM, Kushner FG, Lauer MS, Shaw LJ, Smith SC Jr, Taylor AJ, Weintraub WS, Wenger NK, Jacobs AK, Smith SC Jr, Anderson JL, Albert N, Buller CE, Creager MA, Ettinger SM, Guyton RA, Halperin JL, Hochman JS, Kushner FG, Nishimura R, Ohman EM, Page RL, Stevenson WG, Tarkington LG, Yancy CW; American College of Cardiology Foundation; American Heart Association. 2010 ACCF/AHA guideline for assessment of cardiovascular risk in asymptomatic adults: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2010 Dec 14;56(25):e50-103. doi: 10.1016/j.jacc.2010.09.001. No abstract available. PMID 21144964
- [Result] Nasir K, Michos ED, Blumenthal RS, Raggi P. Detection of high-risk young adults and women by coronary calcium and National Cholesterol Education Program Panel III guidelines. J Am Coll Cardiol. 2005 Nov 15;46(10):1931-6. doi: 10.1016/j.jacc.2005.07.052. Epub 2005 Oct 20. PMID 16286182
- [Result] Akosah KO, Schaper A, Cogbill C, Schoenfeld P. Preventing myocardial infarction in the young adult in the first place: how do the National Cholesterol Education Panel III guidelines perform? J Am Coll Cardiol. 2003 May 7;41(9):1475-9. doi: 10.1016/s0735-1097(03)00187-6. PMID 12742284
- [Result] Kappagoda CT, Amsterdam EA. Assessment of risk for developing coronary heart disease in asymptomatic individuals. J Cardiopulm Rehabil Prev. 2009 Jul-Aug;29(4):207-19. doi: 10.1097/HCR.0b013e3181af6be5. PMID 19628986
- [Result] O'Rourke RA, Brundage BH, Froelicher VF, Greenland P, Grundy SM, Hachamovitch R, Pohost GM, Shaw LJ, Weintraub WS, Winters WL Jr. American College of Cardiology/American Heart Association Expert Consensus Document on electron-beam computed tomography for the diagnosis and prognosis of coronary artery disease. J Am Coll Cardiol. 2000 Jul;36(1):326-40. doi: 10.1016/s0735-1097(00)00831-7. No abstract available. PMID 10898458
- [Result] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Result] Wang L, Jerosch-Herold M, Jacobs DR Jr, Shahar E, Detrano R, Folsom AR; MESA Study Investigators. Coronary artery calcification and myocardial perfusion in asymptomatic adults: the MESA (Multi-Ethnic Study of Atherosclerosis). J Am Coll Cardiol. 2006 Sep 5;48(5):1018-26. doi: 10.1016/j.jacc.2006.04.089. Epub 2006 Aug 17. PMID 16949496
- [Result] Myerburg RJ, Interian A Jr, Mitrani RM, Kessler KM, Castellanos A. Frequency of sudden cardiac death and profiles of risk. Am J Cardiol. 1997 Sep 11;80(5B):10F-19F. doi: 10.1016/s0002-9149(97)00477-3. PMID 9291445
- [Result] Raggi P, Callister TQ, Cooil B, He ZX, Lippolis NJ, Russo DJ, Zelinger A, Mahmarian JJ. Identification of patients at increased risk of first unheralded acute myocardial infarction by electron-beam computed tomography. Circulation. 2000 Feb 29;101(8):850-5. doi: 10.1161/01.cir.101.8.850. PMID 10694523
- [Result] Raggi P, Cooil B, Callister TQ. Use of electron beam tomography data to develop models for prediction of hard coronary events. Am Heart J. 2001 Mar;141(3):375-82. doi: 10.1067/mhj.2001.113220. PMID 11231434
- [Result] Goldstein JA, Chinnaiyan KM, Abidov A, Achenbach S, Berman DS, Hayes SW, Hoffmann U, Lesser JR, Mikati IA, O'Neil BJ, Shaw LJ, Shen MY, Valeti US, Raff GL; CT-STAT Investigators. The CT-STAT (Coronary Computed Tomographic Angiography for Systematic Triage of Acute Chest Pain Patients to Treatment) trial. J Am Coll Cardiol. 2011 Sep 27;58(14):1414-22. doi: 10.1016/j.jacc.2011.03.068. PMID 21939822
- [Result] Cheng VY, Lepor NE, Madyoon H, Eshaghian S, Naraghi AL, Shah PK. Presence and severity of noncalcified coronary plaque on 64-slice computed tomographic coronary angiography in patients with zero and low coronary artery calcium. Am J Cardiol. 2007 May 1;99(9):1183-6. doi: 10.1016/j.amjcard.2006.12.026. Epub 2007 Mar 15. PMID 17478137
- [Result] Gurbel PA, Erlinge D, Ohman EM, Neely B, Neely M, Goodman SG, Huber K, Chan MY, Cornel JH, Brown E, Zhou C, Jakubowski JA, White HD, Fox KA, Prabhakaran D, Armstrong PW, Tantry US, Roe MT; TRILOGY ACS Platelet Function Substudy Investigators. Platelet function during extended prasugrel and clopidogrel therapy for patients with ACS treated without revascularization: the TRILOGY ACS platelet function substudy. JAMA. 2012 Nov 7;308(17):1785-94. doi: 10.1001/jama.2012.17312. PMID 23117779
- [Result] Price MJ, Berger PB, Teirstein PS, Tanguay JF, Angiolillo DJ, Spriggs D, Puri S, Robbins M, Garratt KN, Bertrand OF, Stillabower ME, Aragon JR, Kandzari DE, Stinis CT, Lee MS, Manoukian SV, Cannon CP, Schork NJ, Topol EJ; GRAVITAS Investigators. Standard- vs high-dose clopidogrel based on platelet function testing after percutaneous coronary intervention: the GRAVITAS randomized trial. JAMA. 2011 Mar 16;305(11):1097-105. doi: 10.1001/jama.2011.290. PMID 21406646
- [Result] Collet JP, Cuisset T, Range G, Cayla G, Elhadad S, Pouillot C, Henry P, Motreff P, Carrie D, Boueri Z, Belle L, Van Belle E, Rousseau H, Aubry P, Monsegu J, Sabouret P, O'Connor SA, Abtan J, Kerneis M, Saint-Etienne C, Barthelemy O, Beygui F, Silvain J, Vicaut E, Montalescot G; ARCTIC Investigators. Bedside monitoring to adjust antiplatelet therapy for coronary stenting. N Engl J Med. 2012 Nov 29;367(22):2100-9. doi: 10.1056/NEJMoa1209979. Epub 2012 Nov 4. PMID 23121439
- [Result] Tantry US, Bonello L, Aradi D, Price MJ, Jeong YH, Angiolillo DJ, Stone GW, Curzen N, Geisler T, Ten Berg J, Kirtane A, Siller-Matula J, Mahla E, Becker RC, Bhatt DL, Waksman R, Rao SV, Alexopoulos D, Marcucci R, Reny JL, Trenk D, Sibbing D, Gurbel PA; Working Group on On-Treatment Platelet Reactivity. Consensus and update on the definition of on-treatment platelet reactivity to adenosine diphosphate associated with ischemia and bleeding. J Am Coll Cardiol. 2013 Dec 17;62(24):2261-73. doi: 10.1016/j.jacc.2013.07.101. Epub 2013 Sep 27. PMID 24076493
- [Result] Kuvin JT, Patel AR, Sliney KA, Pandian NG, Sheffy J, Schnall RP, Karas RH, Udelson JE. Assessment of peripheral vascular endothelial function with finger arterial pulse wave amplitude. Am Heart J. 2003 Jul;146(1):168-74. doi: 10.1016/S0002-8703(03)00094-2. PMID 12851627
- [Result] Hamburg NM, Benjamin EJ. Assessment of endothelial function using digital pulse amplitude tonometry. Trends Cardiovasc Med. 2009 Jan;19(1):6-11. doi: 10.1016/j.tcm.2009.03.001. PMID 19467447